CLINICAL TRIAL: NCT00738595
Title: Phase II Multicentre, Randomised, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Effectiveness of EVT 302 in Smoking Cessation, Effect on it Own and in Combination With Open Label Nicotine Replacement Therapy.
Brief Title: Phase II Study to Evaluate the Effectiveness of EVT 302 in Smoking Cessation.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evotec Neurosciences GmbH (Industry)
Collaborators: PRA Health Sciences (Industry); Clinpharm International Management Holding GmbH (Unknown)
Responsible Party: Dr S P Jones, VP Clinical Development, Evotec
Organization: Evotec International GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVT 302/3009; EUDRACT No.: 2008-002472-99
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — sembragiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): EVT 302, 5 mg once Daily
  Interventions: Drug: EVT 302
- 2 (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo
- 3 (Experimental): EVT 302 plus open label Nicotine replacement
  Interventions: Drug: EVT 302 plus open label Nicotine replacement
- 4 (Active Comparator): Placebo plus nicotine replacement therapy
  Interventions: Drug: Placebo plus open label Nicotine Replacement

INTERVENTIONS:
Drug: EVT 302 — EVT 302 5 mg once daily
  Arms: 1
Drug: Placebo — Placebo to match EVT 302, 5 mg
  Arms: 2
Drug: EVT 302 plus open label Nicotine replacement — Double-blind EVT 302 plus open label nicotine replacement
  Arms: 3
Drug: Placebo plus open label Nicotine Replacement — Double-blind placebo plus open label Nicotine replacement patch 21 mg once daily.
  Arms: 4

SUMMARY:
This study will investigate the efficacy of EVT 302, a potent and selective inhibitor of Monoamine Oxidase - B, in improving quit rates in chronic cigarette smokers who are motivated to quit smoking. EVT 302 will be compared to placebo both with and without open label nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Smoker of at least 10 cigarettes daily
* Motivated to quit smoking
* Reports at least one unsuccessful attempt to quit in the last 2 years
* In generally good health
* Provides written informed consent to participate in the sudy

Exclusion Criteria:

* Pregnant or nursing females.
* Women of child-bearing potential must agree to use acceptable contraceptive precautions (contraceptive pill and one barrier method)during the study and for 2-months thereafter
* History of anaphylaxis
* History of alcohol or drug abuse
* History of or current significant medical or psychiatric disorder
* History or presence of cataract or abnormality identified by slit lamp investigation
* Use of other MAO inhibitors, pethidine, SSRIs, tricyclic antidepressants,nasal or oral decongestants or cold medicines containing ephedrine, pseudoephedrine or other sympathomimetics.
* Any medicine contraindicated for use with MAO inhibitors.
* Have or be a carrier of hepatitis B or c or HIV 1 or 2
* Use of tobacco products other than cigarettes
* Use of nicotine replacement therapy in the past month
* Received an investigational drug in the past 30 days
* Previous participation in a study with a MAO-B inhibitor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The four-week continuous quit rate over the last four weeks of treatment | Last 4 weeks of therapy

SECONDARY OUTCOMES:
7 -week abstinence | 7 weeks post quit day
7-day point prevalence quit rate | weekly for 7 weeks
Daily cigarettes smoked | Daily
Change from baseline in the number of cigarettes smoked | Week 8
Minnesota Nicotine Withdrawal Scale | Weekly
Brief Questionnaire of Smoking Urges | Weekly
Modified Cigarette Evaluation Questionnaire | Weekly
Adverse Events | Weekly
Laboratory investigations (Haematology & biochemistry) | Weekly
ECGs | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: H D Stahl, MD, PhD, Principal Investigator — ClinPharm International, Leipzig, Germany
Locations (9):
- Germany (9):
  - Evotec Study Site 2, Berlin
  - Evotec Study Site 3, Bochum
  - Evotec Study Site 8, Chemnitz
  - Evotec Study Site 4, Dresden
  - Evotec Study Site 5, Frankfurt
  - Evotec Study Site 7, Görlitz
  - Evotec Study Site 1, Leipzig
  - Evotec Study Site 6, Magdeburg
  - Evotec Study Site 9, Potsdam

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961